CLINICAL TRIAL: NCT04014621
Title: A Multicenter, Randomized, Double Blind, Sham Controlled Trial to Assess the Efficacy of the Ischemic Stroke System (ISS) in Preventing Progressive Reduction of Salvageable Brain Tissue Volume in Subjects With Acute Ischemic Stroke
Brief Title: Augmenting Cerebral Blood Flow to Preserve the Penumbra Trial
Acronym: ImpACT-P
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: BrainsGate (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLP0050615
Record Dates: First submitted 2018-10-28; First posted 2019-07-10 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Ischemic Stroke
Keywords: acute ischemic stroke; randomized clinical trial; anterior circulation; penumbra
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treated (Active Comparator): Treated arm patients will be implanted and treated with one session of SPG stimulation for 6 hours and 5 additional consecutive sessions (4 hours each) of SPG stimulation, the first starting within 18-24 hours from stroke onset and the others 18-26 hours from previous treatment initiation.
  Interventions: Device: SPG stimulation
- Control (Sham Comparator): Control arm patients will be implanted and receive 6 hours of sham stimulation and 5 additional consecutive sessions (4 hours each) of sham stimulation, the first starting within 18-24 hours from stroke onset and the others 18-26 hours from previous treatment initiation.
  Interventions: Device: SPG stimulation

INTERVENTIONS:
Device: SPG stimulation — The BrainsGate Ischemic Stroke System (ISS) consists of an implantable neurostimulator designed to deliver electrical stimulation to the sphenopalatine ganglion (SPG) and/or nerves within the greater palatine canal and pterygopalatine fossa.

SUMMARY:
The primary objective of the study is to demonstrate that SPG (Sphenopalatine Ganglion) stimulation started within 6 hours from stroke onset slows the expansion of the infarct core volume in acute ischemic stroke.

DETAILED DESCRIPTION:
The goal of this study is to identify Acute Ischemic Stroke patients who have a potentially salvageable penumbra and to test if 6 hours of SPG (Sphenopalatine Ganglion) stimulation may "freeze" the volume of the penumbra and reduce the extent of tissue death.

Following a minimally-invasive implantation of the ISS injectable implant, patients will be randomized to either the Treated or Control arm in a 1:1 ratio. Randomization will be dynamic according to the patient's baseline covariates of core volume, total volume, Hypoperfusion Intensity Ratio (HIR), time to baseline imaging, age, NIHSS. Patients in the Treated arm will be treated with active SPG stimulation while patients in the Control arm will undergo sham treatment. After treatment/sham treatment, patients in both groups will undergo a follow up brain non-contrast CT, CT perfusion and CT angiography imaging, 6:45hrs±15min after baseline CTP initiation.

In the case the patient is cooperative, hand strength (pinch and grasp) evaluations should be assessed before and during the 1st treatment/ sham SPG stimulation session.

Following the assessment of the penumbra (after 6 hours) patients will be treated or sham treated for 5 additional consecutive sessions (4 hours each), the first starting within 18-24 hours from stroke onset and the others 18-26 hours from previous treatment initiation and will be followed for 90 days to assess their clinical outcome. In one session (preferably at day 2) Common Carotid Doppler examination is performed to evaluate blood flow dynamics before and during the treatment/sham session.

After the last treatment session, the implant is removed.

ELIGIBILITY:
Inclusion Criteria:

1. Signs & symptoms consistent with the diagnosis of large vessel occlusion in the anterior circulation
2. Age 18-90 years
3. Baseline NIHSS ≥ 10
4. Ability to initiate treatment within 6 hours from stroke onset. Stroke onset is defined as the time the patient was last seen well.
5. Large vessel total occlusion by CTA
6. Penumbra ≥ 50ml (Difference between Tmax6 volume and the ischemic core volume (CBF<38% volume)
7. Mismatch (Tmax6 volume/ischemic core volume (CBF<38% volume) ≥1.5
8. Core and HIR (Tmax10 / Tmax6) volumes: 1. HIR ≥ 0.5 or 2. 0.35 ≤ HIR < 0.5 and "core volume/time from onset to imaging" ≥ 7mililiter/hour
9. Signed informed consent from patient him/herself or legally authorized representative.

Exclusion Criteria:

1. Unable to undergo a contrast brain perfusion scan, including an allergy to contrast media
2. Opportunity for reperfusion therapy (IV thrombolysis or endovascular treatment)
3. Neuro-imaging evidence of any intracranial hemorrhage or hemorrhagic transformation of brain infarct or other significant abnormality (e.g. tumor, abscess, suspect for subarachnoid hemorrhage, arteriovenous malformation, cerebral aneurysm).
4. Significant mass effect with midline shift.
5. Infarct core volume >150 milliliter
6. Old non-lacunar infarct in the anterior circulation on the ipsilateral hemisphere.
7. Previous stroke in the last 6 months or previous stroke with existing sequelae or with mRS > 0 for any reason
8. Pre-existing Modified Rankin Score >1, even if not stroke-related.
9. Acute symptomatic arterial occlusions in more than one vascular territory confirmed on CTA/MRA (e.g., bilateral MCA occlusions, or an MCA and a basilar artery occlusion).
10. Seizures at stroke onset
11. Baseline blood glucose of <50mg/dL (2.78 mmol) or >400mg/dL (22.20 mmol)
12. Severe, sustained hypertension (Systolic BP >185 mmHg or Diastolic BP >110 mmHg)
13. Current participation in another investigational drug or device study
14. Presumed septic embolus; suspicion of bacterial endocarditis
15. Clinical signs and symptoms or evidence for a relevant lesion by neuro-imaging of an acute ischemic stroke in the posterior circulation (Vertebral, Basilar and/or Posterior Cerebral Artery territories), including but not limited to brain-stem findings and/or cerebellar findings and/or isolated homonymous hemianopia or cortical blindness.
16. Patients with bleeding propensity and/or one of the following: INR > 1.8, prolonged activated partial thromboplastin time (aPTT) ≥ 45 sec., platelets count < 75×10^9/L.
17. Serious systemic infection.
18. Women known to be pregnant or having a positive or indeterminate pregnancy test.
19. Patients with other implanted neural stimulator/ electronic devices (pacemakers).
20. History of SPG ablation ipsilateral to the stroke side.
21. Any condition in the oral cavity that prevents implantation of the INS.
22. Known sensitivity to any medications to be used during study.
23. Subjects who have a clinically significant or unstable medical or surgical condition that may preclude safe and complete study participation. Conditions may include: cardiovascular, vascular, pulmonary, hepatic, renal or neurological (other than acute ischemic stroke), or neoplastic diseases, as determined by medical history, physical examination, laboratory tests, or ECG.
24. Subjects who, in the judgment of the investigator, are likely to be non-compliant or uncooperative during the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-10-20 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Volume of core expansion | Day 1
  The primary outcome measure is the volume of core expansion (in milliliters) in 6:45h±15 min. Core expansion is the difference of two volumes: Core volume (CBF<38%) in follow up CTP (at 6:45h±15 min) and Core volume (CBF<38%) in baseline CTP.
  The difference in the mean core expansion between the Treated and Control groups will be assessed as a continuous variable with adjustment for baseline covariates (Core volume, Total volume, HIR, Time to baseline imaging).
  The two-sided significance level is 0.05.
  Handling of missing data in the primary analysis:
  Patients who die before the 6:45h±15 min follow-up imaging will be assigned a final core volume that equal the baseline total volume.
  Patients with non-interpretable follow-up imaging will be excluded from the analysis.

SECONDARY OUTCOMES:
Difference in infarct volume between baseline CTP core volume and follow up NCCT infarct volume. | Day 1
  Difference in infarct volume (in milliliters) between baseline CTP core volume (CBF<38%) and follow up 6:45h±15 min NCCT infarct volume, adjusted using stratification parameters (Core volume, Total volume, HIR, Time to baseline imaging).
Difference in infarct volume between baseline CTP core volume and Day-5 NCCT infarct volume | Day 5
  Difference in infarct volume (in milliliters) between baseline CTP core volume (CBF<38%) and Day-5 NCCT infarct volume, adjusted using stratification parameters (Core volume, Total volume, HIR, Time to baseline imaging).
3 months mRS | Day 90±7
  mRS at 90-day:
  1. Utility weighted mRS
  2. mRS Dichotomy 0-2
  3. mRS Dichotomy 0-3
Increased blood flow in Common Carotid Doppler | Day 2-6
  Increased blood flow in Common Carotid Doppler (if available).
Improvement in hand motor performance | Day 1
  Improvement in hand motor performance (if available) using a hand dynamometer (Baseline Hydraulic Hand Dynamometers, Fabrication Enterprises Inc, White Plains NY, USA).

OTHER OUTCOMES:
Safety Data Between the Treatment and Control Arms - Serious Adverse Events | Day 90±7
  Incidence of Serious Adverse Events
Safety Data Between the Treatment and Control Arms - Mortality | Day 90±7
  Incidence of Mortality
Safety Data Between the Treatment and Control Arms - Symptomatic Intracranial hemorrhage (sICH) SAEs | Day 5
  Incidence of symptomatic intracranial hemorrhage (sICH) SAEs
Safety Data Between the Treatment and Control Arms - Pain | Day 1 to 5
  Incidence of Pain adverse events during stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Yoram Slolberg, Dr., Study Director — BrainsGate
Locations (4):
- Georgia (4):
  - Academian Z.Tskhakaia West Georgia National Center of Interventional Medicine, Kutaisi
  - Rustavi Central Hospital, Rustavi
  - K. Eristavi National center of clinical and experimental surgery's hospital "New Life", Tbilisi
  - LTD High Technology Medical Center University Clinic, Tbilisi

IPD SHARING:
Plan to Share IPD: No